CLINICAL TRIAL: NCT03376880
Title: Respiratory Effects of Obesity in Children
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tony Babb, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 052012-076
Record Dates: First submitted 2017-07-26; First posted 2017-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Obese Boys: Obese boys group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI > 95th percentile, which will be expressed as a percentage above the 95th percentile < 150% of the 95th percentile.
  Interventions: Other: 1 year follow-up testing
- Obese Girls: Obese girls group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI > 95th percentile, which will be expressed as a percentage above the 95th percentile < 150% of the 95th percentile.
  Interventions: Other: 1 year follow-up testing
- Normal Weight Boys: Normal weight boys group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI between 16th and 84th percentile.
  Interventions: Other: 1 year follow-up testing
- Normal Weight Girls: Normal weight girls group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI between 16th and 84th percentile.
  Interventions: Other: 1 year follow-up testing
- Obese Boys Misdiagnosed with Asthma: Obese boys group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI > 95th percentile, which will be expressed as a percentage above the 95th percentile < 150% of the 95th percentile.This group will have a prior diagnosis of asthma without confirmation by lung function testing.The absence of asthma will be confirmed by a negative response (<10% increase in FEV1) to spirometry before and after bronchodilator (and on visit 2 by a negative bronchial challenge test [<10% decrease in FEV1]; i.e., EVH).
  Interventions: Other: 1 year follow-up testing
- Obese Girls Misdiagnosed with Asthma: Obese girls group defined by a Tanner score ≤ 3 in 8-12 yr olds with a BMI > 95th percentile, which will be expressed as a percentage above the 95th percentile < 150% of the 95th percentile.This group will have a prior diagnosis of asthma without confirmation by lung function testing.The absence of asthma will be confirmed by a negative response (<10% increase in FEV1) to spirometry before and after bronchodilator (and on visit 2 by a negative bronchial challenge test [<10% decrease in FEV1]; i.e., EVH).
  Interventions: Other: 1 year follow-up testing

INTERVENTIONS:
Other: 1 year follow-up testing — The approach of the study is not in studying the effectiveness of the intervention stimulus, the dose response of diet and exercise, or the rate of weight loss but only the response to 1) weight loss and regular exercise or 2) continued weight gain.

SUMMARY:
In obese children, excess fat on the thorax exerts an unfavorable burden on the respiratory system, particularly during exercise; however, it is unclear if this burden reduces exercise tolerance, provokes dyspnea on exertion, or contributes to respiratory symptoms that could be misdiagnosed as asthma, placing obese children at risk of unnecessary treatment and potentially a reluctance to exercise explaining reports of low physical activity and fitness levels, which are counterproductive to weight loss. The investigators will examine the respiratory effects of obesity in prepubescent boys and girls, including those with respiratory symptoms misdiagnosed as asthma, before and after 1) a program of weight loss and regular exercise and 2) continued weight gain as compared with prepubescent normal weight boys and girls before and after 1 year. These results will have broad and immediate clinical impact on the care of obese children, especially those with respiratory symptoms misdiagnosed as asthma, and the results could alter interventional approaches for preventing and treating childhood obesity.

DETAILED DESCRIPTION:
In obese children, excess fat exerts an unfavorable burden on the respiratory system, particularly during exercise, potentially reducing exercise tolerance and leading to DOE (dyspnea on exertion), which could explain reports of low physical activity and fitness levels in obese children. The investigators propose that most of the respiratory effects in obese children are the result of low lung volume breathing, i.e., a reduction in functional residual capacity (FRC) at rest, and end-expiratory lung volume (EELV) during exercise.

The overall objective of this application is to investigate the respiratory effects of obesity in prepubescent children, including obese children with respiratory symptoms misdiagnosed as asthma, before and after 1) a program of weight loss and regular exercise and 2) continued weight gain as compared with normal weight children before and after 1 yr. The investigative approach will be to examine respiratory function, exercise tolerance, and dyspnea on exertion (DOE) in prepubescent obese boys and girls, including those misdiagnosed with asthma (i.e., asthma not confirmed by lung function tests), before and after 1) weight loss (or an equivalent reduction in BMI percentile) and regular exercise and 2) continued weight gain (or an increase in BMI percentile) as compared with prepubescent normal weight boys and girls before and after a control period of 1 yr.

Specific Aims: The following hypotheses will be tested in obese children as compared with normal weight children:

Aim 1) Obesity will decrease respiratory function but to a greater extent in obese children misdiagnosed with asthma as evidenced by altered pulmonary function and breathing mechanics at rest; Aim 2) Obesity will decrease exercise tolerance (as evidenced by peak maximum oxygen uptake (VO2) in ml/min/kg, i.e., physical fitness), but not cardiorespiratory fitness (as evidenced by peak VO2 in % of predicted based on ideal body wt), except in obese children misdiagnosed with asthma where both may be reduced during graded cycle ergometry; Aim 3) Obesity will increase DOE but to a greater extent in obese children misdiagnosed with asthma as evidenced by increased ratings of perceived breathlessness during constant load exercise cycling; and Aim 4) Weight loss and regular exercise will improve respiratory function, exercise tolerance, and DOE in obese children, including those misdiagnosed with asthma, while continued weight gain will worsen respiratory function, exercise tolerance, and DOE in obese children, including those misdiagnosed with asthma, as compared with normal weight children before and after 1 yr.

The long-term objective is to investigate the effects of obesity on respiratory function, exercise tolerance, and DOE, examine obesity-related respiratory symptoms misdiagnosed as asthma in obese children, and provide novel results that could alter interventional approaches for preventing obesity and treating obesity in obese children. Thus, these results will have broad and immediate clinical impact on the care of obese children, especially those with respiratory symptoms misdiagnosed as asthma.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy with normal lung function; prepubescent (Tanner equal to or less than 3); age and gender specific BMI > 95th percentile, but less than 150% of the 95th percentile based on the CDC standards or age and gender specific BMI between the 16th and 84th percentile based on the Center for Disease Control (CDC) standards; and ability to perform pulmonary and exercise test accurately.

Exclusion Criteria:

* Children with significant diseases other than obesity or shortness of breath on exertion will be excluded. Subjects participating in regular conditioning-type vigorous exercise two times or more per week will be excluded (i.e., sports training). Children who are non-English speaking will be excluded from the study because the tests performed are very effort dependent, detailed, and require technical communication between the staff and the child.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants included in the study will be prepubescent boys and girls aged 8-12 yr old of all racial and ethnic origins with a Tanner Pubertal Stage of ≤ 3, and the ability to perform pulmonary function and exercise test accurately.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function: Lung Volumes | Change from Baseline in difference between nonobese and obese children at 1 yr
  Pulmonary function is comprised of several physiological variables but this study will primarily measure Lung Volume: FRC (liters) and TLC (liters)
Exercise Tolerance - Peak VO2 | Change from Baseline differences between nonobese and obese children at 1 yr
  Exercise Tolerances is represented by several physiological variables but the primary variable is Maximal oxygen uptake (L/min and percent predicted)
Dyspnea on Exertion | Change from Baseline differences between nonobese and obese children at 1 yr
  Dyspnea on Exertion is represented using the Borg Scale which provides Ratings of Perceived Breathlessness (RPB) during constant load exercise cycling. The Borg Scale measures from 0-10, where 0 = no breathlessness and 10 = maximal breathlessness.

OTHER OUTCOMES:
Pulmonary Function: Spirometry | Change from Baseline differences between nonobese and obese children at 1 yr
  Spirometry includes: Forced vital capacity (FVC) (liters), Forced Expiratory Volume in 1 second (FEV1) (liters), FEV1/FVC (% ratio), and peak flow (liters/sec)
Pulmonary Function: Diffusing Capacity | Change from Baseline differences between nonobese and obese children at 1 yr
  Diffusing Capacity: Diffusing capacity of lung for carbon monoxide(DLco) (ml/mmHg/min)
Exercise Tolerance: Work Rate | Change from Baseline differences between nonobese and obese children at 1 yr
  Associated variables such as work rate (W)
Exercise Tolerance: Minute Ventilation | Change from Baseline differences between nonobese and obese children at 1 yr
  Associated variables such as pulmonary ventilation (L/min)
Exercise Tolerance: Operational Lung Volumes | Change from Baseline differences between nonobese and obese children at 1 yr
  Associated variables such as operational lung volumes (EELV and EILV as a % of TLC)

CONTACTS AND LOCATIONS:
Overall Officials: Tony G Babb, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine, UT Southwestern and Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03376880/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT03376880/ICF_004.pdf